CLINICAL TRIAL: NCT01119820
Title: Tissue Donation for Myoblast Culture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Felicia Lane, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2008-6467
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Observe in Vitro Characteristics of Muscle Tissue; Elective Obstetric or Gynecologic Surgery
Keywords: elective obstetric or gynecologic surgery
MeSH Terms: interventions — Tissue and Organ Procurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tissue Donation (Experimental): This study will involve females over 18 who are scheduled to undergo elective surgery. These patients will be screened for participation in this study, which will only involve the collection of discarded tissue.
  Interventions: Other: Tissue Donation

INTERVENTIONS:
Other: Tissue Donation — Females over 18 who are scheduled to undergo elective surgery will have discarded tissue collected.

SUMMARY:
Analyze human skeletal muscle and learn more about the ability of adult muscle to produce myoblasts (young muscle cells).

DETAILED DESCRIPTION:
Study the ability of healthy human skeletal muscle to produce myoblasts, and to determine how many cells would be needed to regenerate a certain section of injured muscle. As part of this research, we hope to gain a better understanding of the effect of age on muscle and how normal skeletal muscle can regenerate itself by producing myoblasts. The information gathered from this study will be specifically used in future research for treating Anal Incontinence.

ELIGIBILITY:
Inclusion Criteria:

- Age: 18 years of age or older Female Patients who are already electing to undergo obstetric or gynecologic surgery (either vaginal or abdominal) for a preexisting condition.

Exclusion Criteria:

- Active systemic or pelvic infections including HIV HBV HCV, STD, PID Patients with tumors, metastatic disease or treated with cytostatics Patients undergoing emergency surgical procedures Unconscious or mentally incapable to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
cell expansion | weekly
  The goal of this pilot study is to obtain small amounts of human skeletal muscle that would normally be discarded during gynecologic surgery and instead conserve this tissue for laboratory analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Lane, MD, Principal Investigator — UCI Medical Center
Locations (1):
- UCI Women's Healthcare, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No